CLINICAL TRIAL: NCT03393455
Title: Evolution of Maternal & Infantile Health Following Parental Refusal of Termination of Pregnancy Despite Such Option Being Allowable by the Centre Pluridisciplinary de Diagnostic Prenatal (Interdisciplinary Center for Prenatal Diagnostics)
Brief Title: Obstetric & Pediatric Evolution Following Parental Refusal for Early Termination of Pregnancy Despite Fetal Risk
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0260
Record Dates: First submitted 2017-10-12; First posted 2018-01-08 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-10

CONDITIONS: Termination of Pregnancy
Keywords: Fetal pathology; Obstetrical outcome; Pediatric outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: not accurate — not accurate

SUMMARY:
More and more parents decide to maintain pregnancy which could have been interrupted because of serious fetal pathologies.

In this observational study, the investigators examine obstetrical and pediatric evolution of these pregnancies, from 2006 to 2016 in Montpellier University Hospital.

ELIGIBILITY:
Inclusion criteria:

- refusal of termination of pregnancy despite serious fetal pathology

Exclusion criteria:

* termination of pregnancy
* termination of pregnancy not accepted by the Interdisciplinary Center for Prenatal Diagnostics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mother and child after refusal of termination of pregnancy despite serious fetal pathology
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Apgar score at 5 minutes | 1 day
  Apgar score at 5 minutes

SECONDARY OUTCOMES:
health status of children | 1 day
  health status of children at 1 year old : alive or dead.

CONTACTS AND LOCATIONS:
Overall Officials: florent FUCHS, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC